CLINICAL TRIAL: NCT00576927
Title: Improving Sleep in Nursing Homes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Patricia C Griffiths, Principal Investigator, Emory University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00000460; R01AG028769 (NIH)
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Deprivation
Keywords: Sleep hygiene; Sleep latency; Elderly sleep; Nursing Home sleep
MeSH Terms: conditions — Sleep Deprivation; Sleep Hygiene | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group1 (Experimental): SHI followed by Active Drug Ramelteon
  Interventions: Drug: Ramelteon
- Group 2 (Placebo Comparator): SHI Followed by Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Subjects demonstrating low sleep efficiencies and prolonged sleep latencies, will be randomly assigned to continue to receive SHI accompanied by either placebo or Ramelteon (8 mg). Matching placebo will be obtained and the medication pre-packaged and ordered based on the randomization results.
  Other Names: Rozerem
  Arms: Group1
Drug: Placebo
  Arms: Group 2

SUMMARY:
Older people living in nursing homes do not sleep very well for many reasons. Sleep disorders such as sleep apnea (when someone briefly stops breathing during sleep), and night time urination, along with the problems caused by the nighttime environment of the nursing home, such as noise and disruptive care routines can all contribute. Poor sleep can lead to other health problems or make existing health problems worse.

This study will evaluate how well a sleep hygiene intervention and a medication for sleep (ramelteon (Rozerem)) work to improve sleep in nursing home residents with poor sleep. Ramelteon is FDA approved and has been tested in older adults living in the community, but not in older adults living in nursing homes. We expect sleep to improve on the study drug along with the sleep hygiene intervention, in comparison to placebo along with the sleep hygiene intervention. Based on adverse events reported in previous samples of older subjects, we expect the study drug to cause few side effects.

DETAILED DESCRIPTION:
This study evaluates how well Ramelteon works by measuring sleep at night and during the day. After consenting and final determination of eligibility, participants will complete a baseline phase to assess usual sleep, as well as daytime alertness and activity , thinking and memory, walking and balance (among those who walk and/or stand), and mood. Sleep at night and during the day will be objectively assessed with wrist actigraphs in all subjects. Approximately half will also receive polysomnography to assess nighttime sleep. Subjects who sleep more than 75% of the time they are in bed will not continue in the study. Subjects that do not have improved sleep with the sleep hygiene program will be randomized to one of two treatment groups - one will receive the active drug along with the sleep hygiene intervention and the other will receive a placebo along with the sleep hygiene intervention. Following randomization, subjects will complete a brief run-in phase and then enter the treatment phase. Assessment of sleep and other measures will be repeated.

The primary hypotheses to be examined in this study are as follows:

Hypothesis 1: Subjects treated with ramelteon in addition to a sleep hygiene (SHI) will have improved sleep latency, and as a consequence, a significant increase in actigraphically measured sleep efficiency, compared to subjects treated with placebo plus a SHI.

Hypothesis 2: Subjects treated with ramelteon in addition to a SHI will sleep less and spend less time in bed during the day, be more engaged in daytime activities, and have better mood than subjects treated with placebo plus a SHI.

Hypothesis 3: Changes in daytime sleep, time in bed during the day, engagement in activities, and mood will be positively correlated with improved sleep efficiency among subjects receiving ramelteon in addition to a SHI.

ELIGIBILITY:
Inclusion Criteria:

* After initial screening and consenting, subjects with a 5-night average baseline sleep efficiency of less than or equal to 75% will be included

Exclusion Criteria:

* Less than 65 yrs old
* Bedbound
* Resided in NH for less than two months
* Patients on Medicare Part A skilled Benefit(anticipated short length stay) - Terminal Illness
* Unstable psychotropic drug regimen (addition, discontinuation, or change of dosage of any psychotropic drug in the prior two weeks) - Use of hypnotic, antihistamine, or benzodiazepine more than once per week during the two weeks before screening
* Use of drugs that could potentially inhibit the metabolism of Ramelteon (ie: fluvoxamine, ketoconazole, fluconazole)
* Use of Drugs that induce the metabolism of Ramelteon (ie: rifampin)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Griffiths, PhD, Principal Investigator — Emory University, School of Medicine, Division of General Medicine and Geriatrics

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were long-stay residents of NHs in the Atlanta area who were > age 65. Potential subjects were initially screened using administrative data and medical record review. Potential subjects who do not meet any of the exclusion criteria after initial screening were approached for informed consent or proxy consent was obtained when applicable.
Pre-assignment Details: Those for whom consent was obtained underwent a clinical assessment and baseline measures . Only subjects with 5-night average sleep latency > 20 minutes and/or sleep efficiency <80% were included . Subjects with severe sleep apnea were excluded and referred to their primary physician. Subjects unable to tolerate the actiwatches were excluded.
Period: Clinical Assessment
Arm/Group | All Subjects
Started | 79
Completed | 43
Not Completed | 36
Not completed — Lack of Efficacy | 24
Not completed — Death | 1
Not completed — Withdrawal by Subject | 10
Not completed — Physician Decision | 1
Period: Baseline
Arm/Group | All Subjects
Started | 43
Completed | 30
Not Completed | 13
Not completed — Physician Decision | 9
Not completed — Medication Change by PCP of subject | 1
Not completed — Withdrawal by Subject | 3
Period: Sleep Hygiene Behavioral Intervention
Arm/Group | All Subjects
Started | 30
Completed | 23
Not Completed | 7
Not completed — Responded to intervention | 4
Not completed — Death | 1
Not completed — Medication Change by PCP for subject | 1
Not completed — Withdrawal by Subject | 1
Period: Sleep Hygiene With the Placebo
Arm/Group | All Subjects
Started | 23
Completed | 22
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Sleep Hygiene With Study Drug
Arm/Group | All Subjects
Started | 22
Completed | 22
Not Completed | 0
Period: Randomization 1:1 Placebo or Active Drug
Arm/Group | All Subjects
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects entered a clinical assessment phase (CAP) after consent, which eliminated 36 subjects. Then 43 subjects entered baseline which excluded 13 subjects. 30 subjects started sleep hygiene intervention, but only 23 subjects completed. 1 more subject withdrew during placebo. Then 22 started drug and those 22 completed randomization.
Groups:
- Ramelteon: 6 Weeks of Sleep Hygiene Intervention (SHI) followed by Placebo Run-in (3 days) then Active Drug (Ramelteon) for those whose sleep did not improve.
- Placebo: 6 Weeks of Sleep Hygiene Intervention (SHI) followed by Placebo Run-in (3 days) then Placebo for those whose sleep did not improve with SHI alone.
- Total: Total of all reporting groups
Arm/Group | Ramelteon | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.9 (6.8) | 85.0 (8.9) | 85.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Secondary Outcome: Sleep Efficiency
Description: % of time asleep holding time in bed constant (averaged over 3-5 nights)
Time Frame: All Assessment Phases, up to one week
Population: Per protocol -- intention to treat - ITT - last carried forward.
Measure: Mean (Standard Deviation); unit: percentage of sleep
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 11 | 11
percentage of sleep | 76.5 (11.8) [300 to 400] | 73.8 (14.9) [300 to 400]

2. Primary Outcome: Number of Participants Meeting Good Sleep Latency Criteria
Description: Sleep Latency Criteria for "Good Latency" measured by behavioral observations conducted every 10-15 minutes after 4pm until 11pm.
  Good latency is described as subject asleep in under 20 minutes on 51% of the nights observed in a week.
Time Frame: All assessment periods, up to one week
Population: 30 subjects enrolled into the behavioral intervention. 4 subjects responded to the sleep hygiene intervention (SHI) arm and completed the study. 3 subjects were excluded for various reasons from the SHI arm. 23 subjects continued onto the placebo/SHI. 1 subject withdrew from that arm. From there,11 subjects received drug and 11 remained on placebo
Measure: Number; unit: participants
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 11 | 11
participants | 7 | 6
Statistical Analysis 1: Comparison: Ramelteon vs Placebo; Test type: Superiority or Other; p = 0.655, Chi-squared — p-value suspect because of sparse cell counts; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.156 to 8.717]

3. Secondary Outcome: Daytime Engagement Status
Description: Trained research technicians observed the subjects behavior during assessment phases every 15 minutes for one full minute. Specific behavioral definitions were employed to record whether the subject was in or out of bed, awake or asleep (eyes closed with no purposeful movement for at least 60 consecutive seconds), actively engaged in an activity (reading, watching television, conversation, a specific group activity, etc), and whether any physical or verbal agitation was noted.
Time Frame: All Assessment Phases, up to one week
Measure: Mean (Standard Deviation); unit: percentage of engaged observations
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 11 | 11
percentage of engaged observations | 54.6 (24.6) | 54.6 (24.6)

4. Other Pre Specified Outcome: Daytime Sleep
Description: As measured by percent of daytime behavioral observations observed asleep
Time Frame: All Assessment Phases, up to one week
Measure: Mean (Standard Deviation); unit: percentage of daytime sleep observations
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 11 | 11
percentage of daytime sleep observations | 19.4 (23.1) | 21.7 (29.0)

ADVERSE EVENTS:
Arm/Group | Ramelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Low power to detect statistically significant effects of the interventions on outcomes; Inability to examine predictors of responsiveness because of the small sample size and the large number of predictors of response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No